CLINICAL TRIAL: NCT00623727
Title: Randomized, Active-controlled, Double-blind, Parallel Design Study to Evaluate the Efficacy and Safety of a Once-a-week Prophylaxis Treatment With BAY79-4980 Compared to Three Times-per-week Prophylaxis With rFVIII-FS in Previously Treated Patients With Severe Hemophilia A
Brief Title: BAY79-4980 Compared to rFVIII-FS in Previously Treated Patients With Severe Hemophilia A
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer HealthCare Pharmaceuticals Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12781; 2007-003718-32 (EudraCT Number)
Record Dates: First submitted 2008-01-09; First posted 2008-02-26 (Estimated); Results first posted 2011-08-17 (Estimated); Last update posted 2013-07-15 (Estimated); Status verified 2013-07

CONDITIONS: Hemophilia A
Keywords: Hemophilia A; FVIII disease; rFVIII
MeSH Terms: conditions — Hemophilia A | interventions — BAY 14-2222

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rFVIII-FS/pegylated liposomes (BAY79-4980) (Experimental): 35 IU/kg body weight of BAY79-4980 1x/week plus 2 dummy injections/week (dummy = rFVIII (recombinant factor VIII)-FS (formulated with sucrose) excipient reconstituted in WFI (sterile water for injection))
  Interventions: Biological: rFVIII-FS/pegylated liposomes (BAY79-4980)
- rFVIII-FS/WFI (BAY14-2222) (Active Comparator): 25 IU/kg body weight of rFVIII-FS 3x/week (employing 1 percent POPC (1-palmitoyl-2-oleoyl-sn-glycero-3-phosphocholine)-alone liposome (rFVIII-FS-POPC) as blinding agent used for first weekly injection and rFVIII-FS in WFI for 2nd and 3rd injection)
  Interventions: Biological: rFVIII-FS/WFI (BAY14-2222)

INTERVENTIONS:
Biological: rFVIII-FS/pegylated liposomes (BAY79-4980) — 35 IU/kg body weight intravenous 1x/week for 52 weeks This arm will be stopped by 30.04.10 the subjects will be offered to change to the active comparator arm
  Arms: rFVIII-FS/pegylated liposomes (BAY79-4980)
Biological: rFVIII-FS/WFI (BAY14-2222) — 25 IU/kg body weight intravenous 3x/week for 52 weeks
  Arms: rFVIII-FS/WFI (BAY14-2222)

SUMMARY:
A study to assess treatment with a new formulation of recombinant factor VIII reconstituted with liposomes (BAY79-4980) to evaluate whether a once-a-week treatment is safe and can prevent bleeds in subjects with severe haemophilia A.

ELIGIBILITY:
Inclusion Criteria:

* Males aged 12 to 70 years
* Subjects with severe hemophilia A (< 1% factor VIII [FVIII]:C)
* Subjects with equal or greater than 150 exposure days (EDs) with any FVIII in total
* Subjects who have been on-demand treatment with a minimum of 1 relevant bleed per month or have been on secondary prophylaxis treatment with not more than a 3x/week schedule
* Subjects with bleeding events and/or treatments during the last 6 months prior to study entry which are documented in the subjects medical records
* Subjects with no measurable inhibitor activity
* Subjects with no history of FVIII inhibitor antibody formation
* Written informed consent by subject and parent / legal representative, if < 18 years

Exclusion Criteria:

* Subjects who are receiving primary prophylaxis
* Subjects on prophylaxis with documented requirements of > 75 IU/kg/week
* Subjects with any other bleeding disease beside hemophilia A (i.e., von Willebrand disease)
* Subjects with abnormal renal function
* Subjects with elevated hepatic transaminases
* Subjects on treatment with immunomodulatory agents within the last 3 months prior to study entry or during the study
* Subjects with known hypersensitivity to the active substance, mouse or hamster protein, liposomes or polyethyleneglycol (PEG)
* Subjects who require any pre-medication for FVIII injections

Ages: 12 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2008-06; Primary Completion 2010-04 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (89):
- United States (20):
  - Orange, California
  - Sacramento, California
  - San Francisco, California
  - Aurora, Colorado
  - New Orleans, Louisiana
  - Boston, Massachusetts
  - Detroit, Michigan
  - East Lansing, Michigan
  - Rochester, Minnesota
  - Kansas City, Missouri
  - Las Vegas, Nevada
  - Albuquerque, New Mexico
  - Buffalo, New York
  - Rochester, New York
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Houston, Texas
  - Milwaukee, Wisconsin
- Argentina (2):
  - Buenos Aires, Ciudad Auton. de Buenos Aires
  - Rosario, Santa Fe Province
- Perth, Western Australia, Australia
- Austria (2):
  - Vienna, Vienna
  - Graz
- Belgium (2):
  - Bruxelles - Brussel
  - Leuven
- Canada (6):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Halifax, Nova Scotia
  - Hamilton, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
- Santiago, Chile
- Zagreb, Croatia
- Århus N, Denmark
- Tallinn, Estonia
- France (8):
  - Besançon
  - Le Kremlin-Bicêtre
  - Lyon
  - Marseille
  - Montpellier
  - Paris
  - Rennes
  - Strasbourg
- Germany (3):
  - Bonn, North Rhine-Westphalia
  - Münster, North Rhine-Westphalia
  - Berlin, State of Berlin
- Tel Litwinsky, Israel
- Italy (5):
  - Catania
  - Florence
  - Milan
  - Napoli
  - Torino
- Lithuania (2):
  - Klaipėda
  - Vilnius
- Netherlands (3):
  - Groningen
  - Nijmegen
  - Utrecht
- New Zealand (2):
  - Auckland
  - Christchurch
- Oslo, Norway
- Poland (5):
  - Gdansk
  - Krakow
  - Lodz
  - Poznan
  - Warsaw
- Romania (3):
  - Timișoara, Timiș County
  - Brasov
  - Bucharest
- Johannesburg, Gauteng, South Africa
- Spain (6):
  - Seville, Andalusia
  - Barcelona, Barcelona
  - Madrid, Madrid
  - Oviedo, Principality of Asturias
  - Santa Cruz de Tenerife, Santa Cruz de Tenerife
  - Valencia, Valencia
- Bern, Switzerland
- Taiwan (2):
  - Changhua
  - Taipei
- Turkey (Türkiye) (3):
  - Adana
  - Antalya
  - Izmir
- United Kingdom (6):
  - Cambridge, Cambridgeshire
  - London, London
  - Manchester, Manchester
  - Cardiff, South Glamorgan
  - Sheffield, South Yorkshire
  - Birmingham

REFERENCES:
- [Result] Di Minno G, Cerbone AM, Coppola A, Cimino E, Di Capua M, Pamparana F, Tufano A, Di Minno MN. Longer-acting factor VIII to overcome limitations in haemophilia management: the PEGylated liposomes formulation issue. Haemophilia. 2010 Jan;16 Suppl 1:2-6. doi: 10.1111/j.1365-2516.2009.02155.x. PMID 20059562
- [Result] Powell J, Martinowitz U, Windyga J, Di Minno G, Hellmann A, Pabinger I, Maas Enriquez M, Schwartz L, Ingerslev J; LipLong Study Investigators. Efficacy and safety of prophylaxis with once-weekly BAY 79-4980 compared with thrice-weekly rFVIII-FS in haemophilia A patients. A randomised, active-controlled, double-blind study. Thromb Haemost. 2012 Nov;108(5):913-22. doi: 10.1160/TH12-03-0188. Epub 2012 Sep 26. PMID 23014711

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Previously treated participants with severe hemophilia A (<1% FVIII (Factor VIII)), who were currently on on-demand or secondary prophylaxis treatment with any FVIII for ≥150 exposure days (ED) with documented bleeds/injections during the last 6 months prior to study entry could participate in the study.
Pre-assignment Details: Of 168 enrolled participants, 25 failed screening.
Period: Double Blind (DB)
Arm/Group | rFVIII-FS/Pegylated Liposomes (BAY79-4980) | rFVIII-FS/WFI (BAY14-2222)
Started | 70 (only 67 participants are applicable for baseline characteristic evaluation) | 73 (only 72 participants are applicable for baseline characteristic evaluation)
Participants Received Treatment | 67 | 72
Completed | 34 | 41
Not Completed | 36 | 32
Not completed — Adverse Event | 1 | 3
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 8 | 2
Not completed — Lack of Efficacy | 2 | 2
Not completed — Termination of the double-blind period | 22 | 21
Not completed — Lost to Follow-up | 1 | 1
Not completed — Protocol Violation | 2 | 2
Period: Open Label Follow-up
Arm/Group | rFVIII-FS/Pegylated Liposomes (BAY79-4980) | rFVIII-FS/WFI (BAY14-2222)
Started | 0 | 26 (13 Participants from each group after DB period terminated entered open label follow up.)
Completed | 0 | 18
Not Completed | 0 | 8
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Study termination | 0 | 6
Not completed — Participant convenience | 0 | 1
Period: Open Label Extension Period
Arm/Group | rFVIII-FS/Pegylated Liposomes (BAY79-4980) | rFVIII-FS/WFI (BAY14-2222)
Started | 20 (10 participants of each group entered open-label extension period after completion of DB study) | 0
Completed | 20 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | rFVIII-FS/Pegylated Liposomes (BAY79-4980) | rFVIII-FS/WFI (BAY14-2222) | Total
Number analyzed (Participants) | 67 | 72 | 139
Age Continuous [Mean (Standard Deviation); unit: years] | 33.0 (11.3) | 34.1 (13.0) | 33.5 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 67 | 72 | 139
target joint [Number; unit: participants] — The presence or absence of target joints (defined as joints with at least 3 bleeds into the same joint within 6 months) was evaluated.
  participants
    Yes | 54 | 56 | 110
    No | 13 | 16 | 29
Previous treatment [Number; unit: participants] — Previous treatment was categorized as prophylaxis versus on demand
  participants
    On demand | 35 | 44 | 79
    Prophylaxis | 32 | 28 | 60

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Less Than 9 Total Bleeds Per Year
Description: Bleeds occurring on the same day were counted as one bleeding event. Bleeds occurring within 72 hours into the same location were also counted as one bleeding event.
Time Frame: up to one year
Population: Per protocol (PP) population
Measure: Number; unit: Percentage of participants
Arm/Group | rFVIII-FS/Pegylated Liposomes (BAY79-4980) | rFVIII-FS/WFI (BAY14-2222)
Number analyzed (Participants) | 63 | 68
Percentage of participants | 38.1 | 72.1

2. Secondary Outcome: Percentage of Participants With Less Than 5 Joint Bleeds Per Year
Description: as for outcome 1
Time Frame: up to one year
Population: PP population
Measure: Number; unit: Percentage of participants
Arm/Group | rFVIII-FS/Pegylated Liposomes (BAY79-4980) | rFVIII-FS/WFI (BAY14-2222)
Number analyzed (Participants) | 63 | 68
Percentage of participants | 38.1 | 63.2

3. Secondary Outcome: Number of Joint Bleeds Per Participant Per Year in Responders
Description: Bleeds occurring on the same day were counted as one bleeding event. Bleeds occurring within 72 hours into the same location were also counted as one bleeding event. Responders were the subjects with less than 9 total bleeds per year
Time Frame: up to one year
Population: PP population in responders
Measure: Median (Full Range); unit: Joint bleeds per year
Arm/Group | rFVIII-FS/Pegylated Liposomes (BAY79-4980) | rFVIII-FS/WFI (BAY14-2222)
Number analyzed (Participants) | 24 | 49
Joint bleeds per year | 2.341 [0.00 to 8.91] | 0.000 [0.00 to 7.59]

4. Other Pre Specified Outcome: Number of Bleeds Per Year
Description: Bleeds occurring on the same day were counted as one bleeding event. Bleeds occurring within 72 hours into the same location were also counted as one bleeding event. Number of bleeds 3 weeks after the first infusion per 12 months
Time Frame: up to one year
Population: PP population
Measure: Median (Full Range); unit: bleeds per year
Arm/Group | rFVIII-FS/Pegylated Liposomes (BAY79-4980) | rFVIII-FS/WFI (BAY14-2222)
Number analyzed (Participants) | 63 | 68
bleeds per year | 9.96 [0.0 to 72.2] | 2.20 [0.0 to 22.8]

5. Other Pre Specified Outcome: Percentage of Bleeds Treated by Various Numbers of Injections
Description: as for outcome 1
Time Frame: up to one year
Population: PP Population
Measure: Number; unit: percentage of bleeds
Arm/Group | rFVIII-FS/Pegylated Liposomes (BAY79-4980) | rFVIII-FS/WFI (BAY14-2222)
Number analyzed (Participants) | 63 | 68
percentage of bleeds
  1-2 injections | 88.5 | 93.0
  1 injection | 73.2 | 81.7
  2 injections | 15.3 | 11.3
  3 injections | 6.5 | 2.3
  >3 injections | 5.0 | 4.7

6. Other Pre Specified Outcome: Total rFVIII Consumption Per Year
Description: Total number of units per kg of study medication (rFVIII) administered to participant for one year. rFVIII is recombinant factor VIII, factor VIII is functional coagulation factor
Time Frame: up to one year
Population: ITT population
Measure: Median (Full Range); unit: IU per kg
Arm/Group | rFVIII-FS/Pegylated Liposomes (BAY79-4980) | rFVIII-FS/WFI (BAY14-2222)
Number analyzed (Participants) | 67 | 72
IU per kg | 2524 [1580 to 11788] | 4378 [3701 to 12789]

7. Other Pre Specified Outcome: Percentage of Participants With Less Than 9 Total Bleeds Per Year in the Open Label Extension Period
Description: as for outcome 1
Time Frame: 6 months after start of open label extension period
Population: Participants who completed open label extension period
Measure: Number; unit: Percentage of participants
Arm/Group | rFVIII-FS/Pegylated Liposomes (BAY79-4980) | rFVIII-FS/WFI (BAY14-2222)
Number analyzed (Participants) | 20 | 0
Percentage of participants | 55.0 |

ADVERSE EVENTS:
Groups:
- rFVIII-FS/Pegylated Liposomes (BAY79-4980) - Double Blind: Reporting Group 1 (RG1): Double Blind Study, 35 IU/kg body weight of BAY79-4980 1x/week plus 2 dummy injections/week (dummy = rFVIII-FS excipient reconstituted in WFI)
- rFVIII-FS/WFI (BAY14-2222) - Double Blind: Reporting group 2 (RG2): Double Blind Study, 25 IU/kg body weight of rFVIII-FS 3x/week (employing 1 percent POPC-alone liposome (rFVIII-FS-POPC) as blinding agent used for first weekly injection and rFVIII-FS in WFI for 2nd and 3rd injection)
- rFVIII-FS/WFI (BAY14-2222) - Follow-up: Reporting group 3 (RG3): Open Label Follow-up, 25 IU/kg body weight of rFVIII-FS 3x/week (employing 1 percent POPC-alone liposome (rFVIII-FS-POPC) as blinding agent used for first weekly injection and rFVIII-FS in WFI for 2nd and 3rd injection)
- rFVIII-FS/Pegylated Liposomes (BAY79-4980) - Extension: Reporting group 4 (RG4): Open Label Extension, 35 IU/kg body weight of BAY79-4980 1x/week plus 2 dummy injections/week (dummy = rFVIII-FS excipient reconstituted in WFI)
Arm/Group | rFVIII-FS/Pegylated Liposomes (BAY79-4980) - Double Blind | rFVIII-FS/WFI (BAY14-2222) - Double Blind | rFVIII-FS/WFI (BAY14-2222) - Follow-up | rFVIII-FS/Pegylated Liposomes (BAY79-4980) - Extension
Serious Adverse Events (participants affected / at risk) | 7/67 | 1/72 | 0/26 | 1/20
Other Adverse Events (participants affected / at risk) | 27/67 | 27/72 | 2/26 | 10/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | rFVIII-FS/Pegylated Liposomes (BAY79-4980) - Double Blind (N=67) | rFVIII-FS/WFI (BAY14-2222) - Double Blind (N=72) | rFVIII-FS/WFI (BAY14-2222) - Follow-up (N=26) | rFVIII-FS/Pegylated Liposomes (BAY79-4980) - Extension (N=20)
Glaucoma (Eye disorders) | 1 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oedema (General disorders) | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0 | 0
Tinea pedis (Infections and infestations) | 1 | 0 | 0 | 0
Varicella (Infections and infestations) | 0 | 0 | 0 | 1
Abnormal weight gain (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | rFVIII-FS/Pegylated Liposomes (BAY79-4980) - Double Blind (N=67) | rFVIII-FS/WFI (BAY14-2222) - Double Blind (N=72) | rFVIII-FS/WFI (BAY14-2222) - Follow-up (N=26) | rFVIII-FS/Pegylated Liposomes (BAY79-4980) - Extension (N=20)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 2 | 0 | 2
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 2 | 0 | 0
Pyrexia (General disorders) | 3 | 3 | 1 | 1
Influenza (Infections and infestations) | 5 | 2 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 10 | 12 | 0 | 6
Varicella (Infections and infestations) | 0 | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Blood amylase increased (Investigations) | 1 | 1 | 0 | 1
Lipase increased (Investigations) | 1 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 5 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 0 | 1
Haemophilic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 6 | 8 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 4 | 0 | 0

LIMITATIONS AND CAVEATS:
The recruitment and double-blind study phase were prematurely terminated after a scheduled interim analysis confirmed overt failure regarding the primary endpoint as judged by the independent Data and Safety Monitoring Board.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bayer will have up to 30/45 days to review publications, and may request an additional publication delay of up to 60 days to allow for filing a Patent Application (if applicable).

No publication of single center data should be done prior of publication if multi -center data.